CLINICAL TRIAL: NCT06828237
Title: Open, Non-comparative Study to Evaluate the Effectiveness and Safety of the Medical Device KOS® S in the Correction of Moderate or Severe Infraorbital Hollowing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quantum Beauty Kozmetik (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TGMQUA/0124/MD
Record Dates: First submitted 2025-02-04; First posted 2025-02-14 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-07

CONDITIONS: Infraorbital Hollowing

STUDY DESIGN:
Intervention Model Description: Medical Device (pre-market effectiveness and safety, class III)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KOS® S (Other): An open, non-comparative, interventional single-armed clinical trial.
  Interventions: Device: KOS® S

INTERVENTIONS:
Device: KOS® S — Delivery of medical device as injection

SUMMARY:
The process of facial aging is a result of intricate alterations occurring at both the microscopic and macroscopic levels, leading to changes in facial volume. The observed alterations can be attributed to the process of bone structure resorption, the influence of gravity, redistribution of subcutaneous fat, and injury to the skin. Dermal fillers are utilized for the purpose of enhancing facial features in accordance with the aesthetic ideals of beauty. These ideals prescribe specific curves, contours, dimensions, and ratios that must be achieved in order to create a face that is generally considered appealing. Additionally, dermal fillers are employed to replenish volumetric dimensions and restore a more youthful appearance to the aging face (Wongprasert et al. 2022).

Over a period of time, the convex shape of the midface region has the potential to undergo a flattening or concave transformation. The contour alterations observed can be attributed to the descent of the malar soft tissue complex from the zygoma and orbital rims in an inferomedial direction, as well as the atrophy of the malar fat pad. The malar groove, also known as the zygomatic hollow, is a linear indentation that traverses the zygoma in a diagonal manner, running parallel to the nasolabial fold.

Dermal fillers have the potential to reinstate midface volume effectively and augment malar features. The malar augmentation technique involves using dermal filler materials that provide enhanced structural support, making it an operation that is classified as advanced within the field of dermal fillers (Small, Hoang 2012).

KOS® S in the dermis regulates water balance, osmotic pressure and ion flow and functions as a sieve, excluding certain molecules, enhancing the extracellular domain of cell surfaces and stabilizes skin structures by electrostatic interactions.

The Research Question of the present study is the following: to collect sufficient clinical data to demonstrate compliance with the General Safety and Performance Requirements of KOS® S when used as intended.

The primary objective of the study is to evaluate the effectiveness of KOS® S in correcting "Moderate" or "Severe" infraorbital hollowing by assessing the response rate using the Allergan Infraorbital Hollows Scale (AIHS) from the baseline (Response is defined as at least 1-point improvement on the AIHS at month 3 after last treatment).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by the subject
* Females and males ≥ 22 years of age
* Has "Moderate" or "Severe" infraorbital hollowing (grade 2 or 3 on the AIHS) on the 5-point AIHS for each eye as assessed by the Evaluating Investigator (i.e., both eyes must qualify but do not need to have the same score)
* Ability to follow study instructions and likely to complete all required visits
* Reliable methods of contraception which result in a low failure rate (i.e. less than 1 % per year) for women of childbearing potential, e.g. implants, injectables, combined oral contraceptives, some intrauterine-devices, sexual abstinence or vasectomized partner) for the entire study duration.

Exclusion Criteria:

1. Has hyperpigmentation in the infraorbital area (does not include dark circles under the eyes, not due to hyperpigmentation).
2. Has ever received permanent facial implants (e.g., polymethylmethacrylate, silicone, polytetrafluoroethylene) anywhere in the face or neck, or is planning to be implanted with any of these products during the study
3. Has ever undergone fat injections above the subnasale or is planning to undergo this procedure during the study
4. Has tattoos, piercings, facial hair (i.e., beard, moustache), or scars that would interfere with visual assessment of the infraorbital hollows
5. Has undergone volume augmentation with semi-permanent dermal fillers (e.g., calcium hydroxyapatite, poly-L-lactic acid) or temporary dermal fillers in the malar area, temples, or around the eyes within 12 months before enrolment or is planning to undergo such treatment during the study
6. Using any new over-the-counter or prescription oral or topical, anti-wrinkle products within 30 days before enrolment or is planning to begin using such products during the study. Subjects who have been on a regimen of such products for at least 30 days are eligible for the study if they intend to continue their regimen throughout the study)
7. Has congenital or acquired deformities of theface, lipodystrophy, or poor nutritional status
8. Has active or recurrent inflammation or infection in either eye
9. History of or active autoimmune disease/immune deficiency
10. Taking medications and/or substances known to increase coagulation time (e.g., aspirin, ibuprofen, or herbal supplements) 10 days prior to treatment
11. Simultaneousness with laser therapy or deep chemical peeling
12. Prone to hypertrophic scars
13. History of allergy to hyaluronic acid or any of the product's components
14. History of allergy to lidocaine or local anaesthesia of amide compounds
15. Known case of porphyria
16. Pregnancy or lactation
17. Have a condition or be in a situation that, in the physician's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
18. Untreated epilepsy
19. Hypersensitivity to gram positive bacterial proteins as hyaluronic acid is produced by Streptococcus type bacteria

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with at least 1-point improvement from baseline on the AIHS | 3 month
  Proportion of subjects with at least 1-point improvement from baseline on the AIHS (Allergan Infraorbital Hollows Scale) at month 3 after the last treatment (response rate).
  Allergan Infraorbital Hollows Scale - from 0 (No visible hollowing or volume loss medially or laterally) to 4 (Defined hollowing extends from medial to lateral canthus, severe volume loss creates a marked step along the lid-cheek junction)

SECONDARY OUTCOMES:
Change in the AIHS from baseline | 1, 3, 6 and 12 months
  Change in the AIHS from baseline at 1, 3, 6 and 12 months after the last treatment.
  Allergan Infraorbital Hollows Scale (AIHS) - from 0 (No visible hollowing or volume loss medially or laterally) to 4 (Defined hollowing extends from medial to lateral canthus, severe volume loss creates a marked step along the lid-cheek junction)
Proportion of participants with at least 1-point improvement from baseline on the AIHS | 1, 6 and 12 months
  Proportion of participants with at least 1-point improvement from baseline on the AIHS at 1, 6 and 12 months after the last treatment (response rates) Allergan Infraorbital Hollows Scale (AIHS) - from 0 (No visible hollowing or volume loss medially or laterally) to 4 (Defined hollowing extends from medial to lateral canthus, severe volume loss creates a marked step along the lid-cheek junction)
Change from baseline in FACE-Q Satisfaction with Eyes | 1, 3, 6 and 12 months
  Change from baseline in FACE-Q Satisfaction with Eyes scores at 1, 3, 6 and 12 months after the last treatment.
  FACE-Q Satisfaction with Eyes scale: from 1 (very dissatisfied) to 4 (very satisfied)
Secondary outcomes | 1, 3, 6 and 12 months
  Proportion of participants having a positive aesthetic evolution on the 5-point Global Aesthetic Improvement Scale (GAIS) evaluated by the physician and subject at 1, 3, 6 and 12 months after the last treatment
Short- and long-term adverse effects | 2 weeks, 6, 12 months
  Short- and long-term adverse effects within 2 weeks of the initial or touch-up treatment and during 6, 12 months after the last treatment of the study course, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Behnam D Bayatani, Study Chair
Locations (1):
- Clinica Beyond Dental, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wongprasert P, Dreiss CA, Murray G. Evaluating hyaluronic acid dermal fillers: A critique of current characterization methods. Dermatol Ther. 2022 Jun;35(6):e15453. doi: 10.1111/dth.15453. Epub 2022 Apr 5. PMID 35293660
- [Background] Attenello NH, Maas CS. Injectable fillers: review of material and properties. Facial Plast Surg. 2015 Feb;31(1):29-34. doi: 10.1055/s-0035-1544924. Epub 2015 Mar 12. PMID 25763894
- [Background] Fabi S, Zoumalan C, Fagien S, Yoelin S, Sartor M, Chawla S. A Prospective, Multicenter, Single-Blind, Randomized, Controlled Study of VYC-15L, a Hyaluronic Acid Filler, in Adults for Correction of Infraorbital Hollowing. Aesthet Surg J. 2021 Oct 15;41(11):NP1675-NP1685. doi: 10.1093/asj/sjab308. PMID 34351386
- See also: Champely, S. (2020). pwr: Basic Functions for Power Analysis. R package version 1.3-0. — https://CRAN.R-project.org/package=pwr